CLINICAL TRIAL: NCT05263349
Title: Dream Analysis in COPD Patients
Acronym: Rêve BPCO
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP220143
Record Dates: First submitted 2022-02-21; First posted 2022-03-02 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Dreams; Sleep
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COPD patients: Arm with patients with respiratory disease in whom we study dreams
  Interventions: Other: Typical Dreams Questionnaire; Other: HAD Questionnaire; Other: Dream Booklet
- healthy subject: Arm with healthy subjects whose dream analysis will be used as a basis to compare them to the dreams of COPD patients and see if the disease (COPD) has an influence on the patients' dreams
  Interventions: Other: Typical Dreams Questionnaire; Other: HAD Questionnaire; Other: Dream Booklet

INTERVENTIONS:
Other: Typical Dreams Questionnaire — Each of the dreams was classified according to its thematic content (e.g., being involved in a chase, flying through the air, falling, being lost, losing one's teeth, drowning) in order to in a chase, flying through the air, falling, being lost, losing teeth, drowning) in order to determine the most determine the most frequent themes emerging from our sample. The instrument used used to carry out this classification is the "Typical Dream Questionnaire" of Zadra and Nielsen (1999), which has been validated with more than 600 patients suffering from sleep disorders and and 1200 adults (Nielsen et al., 1999; 2003).
Other: HAD Questionnaire — The HAD scale is an instrument that screens for anxiety and depressive disorders. It includes 14 items rated from 0 to 3. Seven questions relate to anxiety (total A) and seven others to the depressive dimension (total D).
  two scores (maximum score for each score = 21).
Other: Dream Booklet — The patient is asked to write down in a notebook every morning the description of the dreams made during the night and to comment on it if necessary

SUMMARY:
Sleep is a fundamental period in life. In a previous work, the investigators have shown that COPD patients presented on the EEG figures found in patients with chronic pain: Alpha-Delta. The link between dyspnea and pain is very strong and this Alpha-Delta could, in these COPD patients, be the witness of nocturnal dyspnea.

Although it is not possible in a non-awake patient to evaluate reliably the dyspnea, sleep offers us a window on the emotions and the feeling of the patient: Dreams.

A few studies have shown the link between breathing and dreaming, but none of them has focused on nocturnal dyspnea.

Our working hypothesis is that respiratory abnormalities in COPD patients are responsible for nocturnal dyspnea, which is reflected in the content of these patients' dreams.

DETAILED DESCRIPTION:
Sleep is a fundamental period for maintaining homeostasis and ensuring many vital functions. It is crucial for brain development, memory and the preservation of our cognitive abilities. It is essential for the adjustment of numerous hormonal secretions, for glycemic control and for the efficiency of our immune system. Today, it is assumed that the reduction of sleep time or the alteration of its quality favors weight gain and obesity, the appearance of diabetes or the development of cancerous diseases. This is a major issue for our modern societies

In patients with respiratory diseases, and in particular with chronic obstructive pulmonary disease (COPD), sleep complaints are extremely frequent. Thus, patients with COPD have subjectively and objectively impaired sleep quality with a lower efficiency and a decrease in the amount of deep slow wave sleep. Moreover, the alteration of the quality of sleep and the physiological modifications of the ventilation during it, worsen the respiratory state of these patients, with an increase of the alveolar hypoventilation, an alteration of the quality of life and an increased risk of exacerbation. A preliminary work of our team was interested in the study of this sleep-breathing relationship and its impact in COPD patients.

Twenty-nine COPD patients hospitalized after respiratory exacerbation were examined by polysomnography. The most striking features were the presence of short (median 328 min, IQR25-75 [299-414]) and poor quality sleep (median Efficiency at 66% IQR 28-75 [51-78]). The sleep architecture was extremely disturbed with notably a decrease in the duration of deep slow-wave sleep with 85 minutes of N3 in median, IQR 25-75 [62-111]. In 3 patients, there was even a complete absence of REM sleep (SP). However, these results only confirmed the data in the literature on the study of sleep in COPD patients.

However, this work has allowed us to highlight 2 other anomalies 1- the demonstration of an electromyographic activation of the cervical inspiratory muscles (MIC) (sternocleidomastoid and scalene) in 26 out of 29 patients during sleep. Activation which, for half of the cases, is not present during wakefulness and only appears during sleep. Moreover, this activation was even present during REM sleep in 9 patients, whereas REM sleep is defined by an abolition of muscle tone. 2- The presence of Alpha Delta on the EEG. This phenomenon has already been observed in patients with chronic pain and is, according to the authors, a sign of cortical integration of pain during sleep.

Dyspnea, or "unpleasant breathlessness", is an abnormal and uncomfortable perception of breathing. The experience of dyspnea is the result of multiple interactions between physiological and environmental factors: it is a complex symptom that signals a threat to homeostasis, frequently inducing an adaptive behavioral response, which is not always efficient. It is responsible for a suffering whose mechanisms and perception can be similar to those of pain. Dyspnea is a subjective sensation with a sensory component and an affective component.

Patients suffering from chronic respiratory disease and in particular COPD very frequently present this symptom of dyspnea on awakening. But during the night, several arguments plead for the persistence of this dyspnea: the activation of the accessory muscles at the cervical level is associated with this sensation of dyspnea and the presence of Alpha Delta at the EEG, known to be a sign of pain during sleep, could in this case be a sign of dyspnea, indeed, the mechanisms of the perception of pain and dyspnea are close.

Although it is often studied, especially in intensive care unit with sedated patients, there is no tool to evaluate dyspnea in non-awake patients. However, sleep is not a state similar to coma or sedation. As everyone knows, sleep is accompanied by a unique cognition: dreams. The scientific term dream includes thoughts, images, sounds, sensations or emotions occurring during sleep.

The link between dreams and breathing has already been established in 2 studies. In the first one, Oudiette et al. showed in lucid dreamers an interaction between the content of their dream (Crossing a nauseating city) and breathing (Apnea preceded by a deep inspiration, witnessing a cortical preparation). Carrasco et al. have shown that the quantity of dreams and their content were related to the effectiveness of the treatment in apneic subjects. The investigators can therefore hypothesize that if patients have respiratory abnormalities responsible for nocturnal dyspnea, these could be reflected in their dreams.

COPD is one of the most frequent respiratory pathologies in France and in the world. The WHO forecasts that it will be the 3rd cause of death in 2030. The study of COPD is therefore a priority, and it is one of the chronic diseases referenced by the Ministry of Solidarity and Health in its national health strategy 2018-2022.

In order to have a comparable control group, patients will be matched to a group of healthy subjects of the same sex and age.

The investigators dream all night long but there is still a difference between dream activity in MS and slow wave sleep. Thus, compared to slow wave sleep, dreams reported after waking up in MS are typically longer, more vivid, more animated (more movement), more emotionally charged and less related to waking experiences. In contrast to MS dreams, slow wave sleep dreams are more closely related to "thoughts" or representations of real life problems.

In this work, The investigators will study the dreams of the patients through 2 tools: a questionnaire of typical dreams in order to have an evaluation of the content of the dreams on the life of the patient (Cf Appendix) as well as a dream diary over 2 weeks to try to have a precise description of the dreams of the patients.

There are no studies that have looked at the dreams of COPD patients. However, it seems necessary to carry out a dream diary over several days in order to accustom the patient to remember his dreams and to succeed in telling them. A duration of 2 weeks seems to be an appropriate compromise between a sufficiently long time to allow relevant information to be collected, without being too long and discouraging for the patients.

ELIGIBILITY:
Inclusion Criteria:

* For both groups:
* Age ≥ 18 years
* Able to understand information and express non-opposition.
* Information and non-opposition gathered
* Affiliated with a social security system
* For patients:
* With confirmed COPD prior to hospitalization at the SRH
* Hospitalized at the SSR of the Pitié-Salpêtrière Hospital

Exclusion Criteria:

For both groups:

* Patient under constraint
* Patient who cannot read or write French
* Patient under AME For healthy subjects
* Known respiratory pathology
* Obesity with BMI > 35 kg/m².
* Known sleep apnea syndrome
* Smoking > 30 PA

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with COPD hospitalized in the respiratory and neuro-respiratory follow-up and rehabilitation department (SSR) of the Pitié-Salpêtrière Hospital.
  Healthy subjects without respiratory disorders selected to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-15 (Actual)

PRIMARY OUTCOMES:
Evaluation of the dreams reported by the patient during 15 days | 15 days after inclusion
  analysis of the dream book filled in by the patient during 15 days

SECONDARY OUTCOMES:
Typical Dream Questionnaire | to inclusion
  The typical dream questionnaire asks how many times the patient has dreamed of the 56 themes listed, the most frequent theme, the theme that occurred earlier in his life, how many dreams he often has in 1 month, the number of nightmares he remembers in a month and the level of distress felt in general in relation to his nightmares. The answers to these questions are then analyzed.
HAD Scale | to inclusion
  The HAD scale is an instrument for detecting anxiety and depressive disorders. It has 14 items rated from 0 to 3. Seven questions relate to anxiety (total A) and seven others to depressive dimension (total D), thus allowing the obtaining of two scores (maximum score of each score = 21).

CONTACTS AND LOCATIONS:
Locations (1):
- SSR Respiratory and Neuro Respiratory, Paris, France